CLINICAL TRIAL: NCT00704288
Title: A Phase 2 Study of XL184 in Subjects With Progressive or Recurrent Glioblastoma Multiforme in First or Second Relapse
Brief Title: Study of XL184 (Cabozantinib) in Adults With Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-201
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; Malignant gliomas
MeSH Terms: conditions — Glioblastoma; Glioma

ARMS (3):
- Group A cabozantinib 175 mg (Experimental): cabozantinib, 175 mg, taken orally once per day (qd).
  Interventions: Drug: XL184
- Group B cabozantinib 125 mg (Experimental): cabozantinib, 125 mg, taken orally once per day (qd).
  Interventions: Drug: XL184
- Group C 125 mg (Experimental): cabozantinib, 125 mg, taken orally once per day (qd).
  Interventions: Drug: XL184

INTERVENTIONS:
Drug: XL184 — Gelatin capsules supplied in 25-mg and 100-mg strengths; continuous daily dosing

SUMMARY:
The purpose of this study is to evaluate the objective response rate and 6-month progression-free survival rate of XL184 in subjects with recurrent or progressive glioblastoma multiforme. XL184 is a new chemical entity that inhibits VEGFR2, MET and RET, kinases implicated in tumor formation, growth and migration.

ELIGIBILITY:
Inclusion Criteria:

* The subject has locally determined histologically confirmed diagnosis of Grade 4 astrocytic tumor.
* The subject has received prior standard radiation for Grade 3 or 4 astrocytic tumor.
* The subject has received prior temozolomide therapy for Grade 3 or 4 astrocytic tumor (if in first relapse, the subject must have received temozolomide until progression, intolerance, or completion of planned therapy; if in second relapse, the subject must have received temozolomide until progression, intolerance, or completion of planned therapy either for first-line treatment or for treatment after first relapse).
* The subject is in first or second Grade 4 relapse, defined as having one or two progressions as Grade 4 astrocytic tumor since the original diagnosis of any grade glioma.
* The subject must have a baseline brain MRI scan within 14 days prior to first dose of XL184 while either not receiving glucocorticoids during the 5 days prior to the baseline MRI scan or on a stable dose of glucocorticoids during the 5 days prior to the baseline MRI scan.
* Subjects having undergone recent resection or biopsy of tumor will be eligible as long as all of the following conditions apply: First dose of XL184 occurs at least 28 days after surgery, the subject has recovered from the effects of surgery, and the subject has measurable residual disease.
* The subject is at least 18 years old.
* The subject has a KPS (Karnofsky Performance Scale) of ≥ 70%.
* The subject is capable of understanding the protocol and has signed the informed consent document.
* The subject has adequate organ and marrow function.
* Sexually active subjects (male and female) must agree to use medically accepted methods of contraception during the course of the study and for 3 months following discontinuation of study drug.
* Female subjects of childbearing potential must have a negative pregnancy test at enrollment.

Exclusion Criteria:

* The subject has received non-standard radiation therapy for glioblastoma, non-anti-angiogenic therapy (including investigational agents, small-molecule kinase inhibitors, and biologic agents) or non-cytotoxic hormonal agent within 28 days of the first scheduled dose of XL184 or mitomycin C within 42 days of the first scheduled dose of XL184, other investigational therapy (including agents not specified above) within 28 days of the first scheduled dose of XL184, or prior treatment with nitrosoureas (including carmustine wafer) at any time.
* Some subjects may not have had any prior VEGF- or VEGFR2-based anti-angiogenic therapy (such as bevacizumab, cediranib, or pazopanib).
* Some subjects may not have had bevacizumab within 14 days of the first scheduled dose of XL184.
* The subject is receiving warfarin (or other coumarin derivatives) at study entry and unable to switch to low molecular weight heparin.
* The subject has evidence of acute intracranial or intratumoral hemorrhage either by MRI or computerized tomography (CT) scan. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin may enter the study.
* The subject is unable to undergo MRI scan (eg, has pacemaker).
* The subject has received enzyme-inducing anti-epileptic agents within 2 weeks before the first dose of XL184 (eg, carbamazepine, phenytoin, phenobarbital, primidone).
* The subject has not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Grade ≤ 1 from adverse events (AEs) due to surgery, antineoplastic agents, investigational drugs, or other medications that were administered before study enrollment.
* The subject has evidence of wound dehiscence.
* The subject is pregnant or breast-feeding.
* The subject has serious intercurrent illness, such as uncontrolled hypertension, unhealed wounds from recent surgery or cardiac arrhythmias or a recent history of significant disease such as either symptomatic congestive heart failure or unstable angina pectoris within the past 3 months, myocardial infarction within the past 6 months, or active infection requiring systemic treatment/hospitalization within 2 weeks of the first scheduled dose of XL184
* The subject has inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* The subject has received any live virus vaccine within 28 days or any inactivated vaccine within 7 days prior to first dose of XL184.
* The subject has had another diagnosis of malignancy (unless nonmelanoma skin cancer, in situ carcinoma of the cervix, or a malignancy diagnosed ≥ 2 years previously) or currently has evidence of malignancy (unless non-melanoma skin cancer or in situ carcinoma of the cervix).
* The subject has a known allergy or hypersensitivity to any of the components of the XL184 formulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2008-05; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Duke University, The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Ellingson BM, Hagiwara A, Morris CJ, Cho NS, Oshima S, Sanvito F, Oughourlian TC, Telesca D, Raymond C, Abrey LE, Garcia J, Aftab DT, Hessel C, Rachmilewitz Minei T, Harats D, Nathanson DA, Wen PY, Cloughesy TF. Depth of Radiographic Response and Time to Tumor Regrowth Predicts Overall Survival Following Anti-VEGF Therapy in Recurrent Glioblastoma. Clin Cancer Res. 2023 Oct 13;29(20):4186-4195. doi: 10.1158/1078-0432.CCR-23-1235. PMID 37540556
- [Derived] Ellingson BM, Aftab DT, Schwab GM, Hessel C, Harris RJ, Woodworth DC, Leu K, Chakhoyan A, Raymond C, Drappatz J, de Groot J, Prados MD, Reardon DA, Schiff D, Chamberlain M, Mikkelsen T, Desjardins A, Holland J, Ping J, Weitzman R, Wen PY, Cloughesy TF. Volumetric response quantified using T1 subtraction predicts long-term survival benefit from cabozantinib monotherapy in recurrent glioblastoma. Neuro Oncol. 2018 Sep 3;20(10):1411-1418. doi: 10.1093/neuonc/noy054. PMID 29660005
- [Derived] Cloughesy TF, Drappatz J, de Groot J, Prados MD, Reardon DA, Schiff D, Chamberlain M, Mikkelsen T, Desjardins A, Ping J, Holland J, Weitzman R, Wen PY. Phase II study of cabozantinib in patients with progressive glioblastoma: subset analysis of patients with prior antiangiogenic therapy. Neuro Oncol. 2018 Jan 22;20(2):259-267. doi: 10.1093/neuonc/nox151. PMID 29036345
- [Derived] Wen PY, Drappatz J, de Groot J, Prados MD, Reardon DA, Schiff D, Chamberlain M, Mikkelsen T, Desjardins A, Holland J, Ping J, Weitzman R, Cloughesy TF. Phase II study of cabozantinib in patients with progressive glioblastoma: subset analysis of patients naive to antiangiogenic therapy. Neuro Oncol. 2018 Jan 22;20(2):249-258. doi: 10.1093/neuonc/nox154. PMID 29016998
- [Derived] Ellingson BM, Harris RJ, Woodworth DC, Leu K, Zaw O, Mason WP, Sahebjam S, Abrey LE, Aftab DT, Schwab GM, Hessel C, Lai A, Nghiemphu PL, Pope WB, Wen PY, Cloughesy TF. Baseline pretreatment contrast enhancing tumor volume including central necrosis is a prognostic factor in recurrent glioblastoma: evidence from single and multicenter trials. Neuro Oncol. 2017 Jan;19(1):89-98. doi: 10.1093/neuonc/now187. Epub 2016 Aug 31. PMID 27580889

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group A (175 mg): Cabozantinib 175 mg (L-malate salt weight; 140 mg freebase equivalent) taken orally once per day (qd)
- Treatment Group B (125 mg); Treatment Group C (125 mg): Cabozantinib 125 mg (L-malate salt weight; 100 mg freebase equivalent) taken orally once per day (qd)
Period: Overall Treatment Period
Arm/Group | Treatment Group A (175 mg) | Treatment Group B (125 mg) | Treatment Group C (125 mg)
Started | 46 | 59 | 117
Naïve | 34 | 37 | 81
Pre-treated | 12 | 22 | 36
Completed | 0 | 0 | 0
Not Completed | 46 | 59 | 117
Not completed — Adverse Event | 11 | 8 | 22
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Disease progression--per Modified MacDonald Criteria (Group A) | 30 | 0 | 0
Not completed — Disease Progression--Radiologic Progression (Group B and C) | 0 | 42 | 76
Not completed — Disease Progression--Clinical Deterioration | 3 | 6 | 11
Not completed — Roll-over to another study | 1 | 0 | 4
Not completed — Other--Subject had intracranial hemorrhage | 1 | 0 | 0
Period: Extended Post Treatment Follow Up Period
Arm/Group | Treatment Group A (175 mg) | Treatment Group B (125 mg) | Treatment Group C (125 mg)
Started (Subjects had a Post-Treatment Visit 30 (+7) days after the final dose of cabozantinib for designated assessments. Thereafter, during extended Post-Treatment Follow-up, information was collected quarterly until death or loss to follow-up. All participants that started the study also started the follow-up period except for subjects who deceased during the study treatment period.) | 46 | 59 | 117
Completed (Completed subjects were not discontinued from the extended post treatment follow up. Not completed subjects were discontinued from the extended post treatment follow up.) | 0 | 0 | 0
Not Completed | 46 | 59 | 117
Not completed — Death | 41 | 50 | 93
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Various reasons | 5 | 5 | 21

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group B + Group C (125 mg): Cabozantinib 125 mg (L-malate salt weight; 100 mg freebase equivalent) taken orally once per day (qd)
- Total: Total of all reporting groups
Arm/Group | Treatment Group A (175 mg) | Treatment Group B + Group C (125 mg) | Total
Number analyzed (Participants) | 46 | 176 | 222
Age, Customized [Count of Participants; unit: Participants]
  18 to <45 | 11 | 33 | 44
  45 to <55 | 11 | 53 | 64
  55 to <65 | 18 | 61 | 79
  65 to <75 | 6 | 28 | 34
  >= 75 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 68 | 83
  Male | 31 | 108 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 40 | 158 | 198
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Response and progression were determined per modified MacDonald Criteria and modified RANO criteria for GBM using imaging and clinical features
Time Frame: 8 weeks until progressive disease
Measure: Number; unit: percentage of participants
Groups:
- Treatment Group A1 (175 mg) - Naive; Treatment Group A2 (175 mg) - Pre-Treated: Cabozantinib 175 mg (L-malate salt weight; 140 mg freebase equivalent) taken orally once per day (qd)
- Treatment Group B1 (125 mg) - Naive; Treatment Group C1 (125 mg) - Naive; Treatment Group B2 (125 mg) - Pre-Treated; Treatment Group C2 (125 mg) - Pre-Treated: Cabozantinib 125 mg (L-malate salt weight; 100 mg freebase equivalent) taken orally once per day (qd)
Arm/Group | Treatment Group A1 (175 mg) - Naive | Treatment Group B1 (125 mg) - Naive | Treatment Group C1 (125 mg) - Naive | Treatment Group A2 (175 mg) - Pre-Treated | Treatment Group B2 (125 mg) - Pre-Treated | Treatment Group C2 (125 mg) - Pre-Treated
Number analyzed (Participants) | 34 | 37 | 80 | 12 | 22 | 36
percentage of participants | 17.6 | 27.0 | 8.8 | 8.3 | 0 | 5.6

2. Secondary Outcome: Duration of Objective Response (Months)
Description: Duration of response is defined as the time from the first documentation of objective response that was subsequently confirmed at a visit that was ≥ 28 days later to disease progression or death due to any cause.
Time Frame: Assessed during periodically scheduled visits until progressive disease
Population: Insufficient number of participants with events
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group A1 (175 mg) - Naive | Treatment Group B1 (125 mg) - Naive | Treatment Group C1 (125 mg) - Naive | Treatment Group A2 (175 mg) - Pre-Treated | Treatment Group B2 (125 mg) - Pre-Treated | Treatment Group C2 (125 mg) - Pre-Treated
Number analyzed (Participants) | 6 | 10 | 7 | 1 | 0 | 2
Months | 5.913 [2.760 to 12.812] | 8.541 [3.778 to 9.264] | NA [2.792 to NA] — Median duration of response and its 95% CI upper limit are not estimable due to insufficient number of events and/or follow up | NA [NA to NA] — Insufficient number of participants with events |  | 4.172 [NA to NA] — Insufficient number of participants with events

3. Secondary Outcome: Progression Free Survival (PFS)
Description: as for outcome 1
Time Frame: Assessed during periodically scheduled visits until progressive disease
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Treatment Group A2 (175 mg) - Pre-Treated; Treatment Group B2 (125 mg) - Pre-Treated; Treatment Group C2 (125 mg) - Pre-Treated: Cabozantinib 125 mg (L-malate salt weight; 100 mg freebase equivalent) taken orally once per day (qd)
Arm/Group | Treatment Group A1 (175 mg) - Naive | Treatment Group B1 (125 mg) - Naive | Treatment Group C1 (125 mg) - Naive | Treatment Group A2 (175 mg) - Pre-Treated | Treatment Group B2 (125 mg) - Pre-Treated | Treatment Group C2 (125 mg) - Pre-Treated
Number analyzed (Participants) | 34 | 37 | 81 | 12 | 22 | 36
Months | 3.712 [1.905 to 5.092] | 4.698 [3.647 to 9.231] | 3.712 [2.562 to 3.712] | 3.285 [0.953 to NA] — Insufficient number of participants with events | 1.807 [1.675 to 3.745] | 2.300 [2.201 to 2.464]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from first dose to death due to any cause.
Time Frame: Assessed during periodically scheduled visits until progressive disease
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Treatment Group A (175 mg) - Naive; Treatment Group A (175 mg) - Pre-Treated: Cabozantinib 175 mg (L-malate salt weight; 140 mg freebase equivalent) taken orally once per day (qd)
- Treatment Group B (125 mg) - Naive; Treatment Group B (125 mg) - Pre-Treated; Treatment Group C (125 mg) - Naive; Treatment Group C (125 mg) - Pre-Treated: Cabozantinib 125 mg (L-malate salt weight; 100 mg freebase equivalent) taken orally once per day (qd)
Arm/Group | Treatment Group A (175 mg) - Naive | Treatment Group A (175 mg) - Pre-Treated | Treatment Group B (125 mg) - Naive | Treatment Group B (125 mg) - Pre-Treated | Treatment Group C (125 mg) - Naive | Treatment Group C (125 mg) - Pre-Treated
Number analyzed (Participants) | 34 | 12 | 37 | 22 | 81 | 36
Months | 7.671 [5.913 to 13.502] | 4.074 [1.380 to 16.689] | 10.381 [7.260 to 16.393] | 4.221 [1.971 to 5.716] | 10.217 [8.016 to 12.122] | 4.583 [2.792 to 5.683]

ADVERSE EVENTS:
Arm/Group | Treatment Group A (175 mg) | Treatment Group B + Group C (125 mg)
All-Cause Mortality (participants affected / at risk) | 41/46 | 144/176
Serious Adverse Events (participants affected / at risk) | 24/46 | 90/176
Other Adverse Events (participants affected / at risk) | 46/46 | 176/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group A (175 mg) (N=46) | Treatment Group B + Group C (125 mg) (N=176)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3
Diverticular Perforation (Gastrointestinal disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Disease Progression (General disorders) | 0 | 5
Asthenia (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Chest Pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1 — Reported term is DEATH UNEXPLAINED
Gait Disturbance (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 2
Gastrointestinal Viral Infection (Infections and infestations) | 0 | 1
H1n1 Influenza (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
Herpes Oesophagitis (Infections and infestations) | 1 | 0
Perirectal Abscess (Infections and infestations) | 1 | 0
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 3
Alanine Aminotransferase Increased (Investigations) | 1 | 3
Aspartate Aminotransferase Increased (Investigations) | 0 | 3
Lipase Increased (Investigations) | 1 | 2
Troponin I Increased (Investigations) | 2 | 0
Amylase Increased (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 2
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Intracranial Tumor Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 6 | 13
Hemiparesis (Nervous system disorders) | 0 | 8
Haemorrhage Intracranial (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 0 | 3
Ataxia (Nervous system disorders) | 0 | 2
Grand Mal Convulsion (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 0 | 2
Acquired Epileptic Aphasia (Nervous system disorders) | 0 | 1
Brain Stem Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral Cyst (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Coordination Abnormal (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial Pressure Increased (Nervous system disorders) | 0 | 1
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 1
Nervous System Disorder (Nervous system disorders) | 0 | 1
Pyramidal Tract Syndrome (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 3 | 4
Mental Status Changes (Psychiatric disorders) | 0 | 4
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Acute Prerenal Failure (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 12
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Interstitial Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Craniotomy (Surgical and medical procedures) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 10
Malignant Hypertension (Vascular disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group A (175 mg) (N=46) | Treatment Group B + Group C (125 mg) (N=176)
Fatigue (General disorders) | 35 | 132
Diarrhoea (Gastrointestinal disorders) | 31 | 97
Decreased Appetite (Metabolism and nutrition disorders) | 22 | 66
Nausea (Gastrointestinal disorders) | 17 | 65
Headache (Nervous system disorders) | 20 | 59
Constipation (Gastrointestinal disorders) | 22 | 54
Hypertension (Vascular disorders) | 18 | 56
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 17 | 56
Alanine Aminotransferase Increased (Investigations) | 15 | 54
Aspartate Aminotransferase Increased (Investigations) | 16 | 49
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 | 49
Blood Lactate Dehydrogenase Increased (Investigations) | 11 | 49
Weight Decreased (Investigations) | 13 | 46
Convulsion (Nervous system disorders) | 9 | 35
Confusional State (Psychiatric disorders) | 8 | 42
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 41
Stomatitis (Gastrointestinal disorders) | 17 | 31
Gait Disturbance (General disorders) | 12 | 34
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 41
Vomiting (Gastrointestinal disorders) | 13 | 29
Insomnia (Psychiatric disorders) | 13 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 29
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 9 | 31
Abdominal Pain (Gastrointestinal disorders) | 12 | 27
Memory Impairment (Nervous system disorders) | 8 | 31
Proteinuria (Renal and urinary disorders) | 13 | 26
Rash (Skin and subcutaneous tissue disorders) | 9 | 30
Depression (Psychiatric disorders) | 5 | 33
Lipase Increased (Investigations) | 6 | 30
Anxiety (Psychiatric disorders) | 7 | 29
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 10 | 26
Leukopenia (Blood and lymphatic system disorders) | 1 | 35
Cognitive Disorder (Nervous system disorders) | 9 | 27
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 12 | 23
Oral Pain (Gastrointestinal disorders) | 5 | 29
Dry Skin (Skin and subcutaneous tissue disorders) | 14 | 19
Dysgeusia (Nervous system disorders) | 7 | 26
Dyspepsia (Gastrointestinal disorders) | 6 | 27
Hemiparesis (Nervous system disorders) | 3 | 27
Oedema Peripheral (General disorders) | 7 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 23
Speech Disorder (Nervous system disorders) | 5 | 25
Dizziness (Nervous system disorders) | 12 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 21
Urinary Tract Infection (Infections and infestations) | 9 | 18
Lymphopenia (Blood and lymphatic system disorders) | 10 | 19
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 7 | 20
Neutropenia (Blood and lymphatic system disorders) | 6 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 21
Ataxia (Nervous system disorders) | 3 | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 17
Mucosal Inflammation (General disorders) | 3 | 20
Sinus Bradycardia (Cardiac disorders) | 4 | 19
Agitation (Psychiatric disorders) | 4 | 18
Aphasia (Nervous system disorders) | 6 | 14
Asthenia (General disorders) | 2 | 17
Deep Vein Thrombosis (Vascular disorders) | 2 | 9
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 | 17
Blood Bilirubin Increased (Investigations) | 7 | 11
Dysphagia (Gastrointestinal disorders) | 3 | 16
Nervous System Disorder (Nervous system disorders) | 6 | 12
Dehydration (Metabolism and nutrition disorders) | 4 | 9
Somnolence (Nervous system disorders) | 5 | 12
Urinary Incontinence (Renal and urinary disorders) | 3 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 13
Dry Mouth (Gastrointestinal disorders) | 4 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Hypothyroidism (Endocrine disorders) | 6 | 11
Vision Blurred (Eye disorders) | 7 | 10
Anaemia (Blood and lymphatic system disorders) | 3 | 13
Flatulence (Gastrointestinal disorders) | 3 | 13
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 11
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 10
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 12
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 10
Amylase Increased (Investigations) | 2 | 11
Contusion (Injury, poisoning and procedural complications) | 2 | 11
Dysarthria (Nervous system disorders) | 2 | 11
Faecal Incontinence (Gastrointestinal disorders) | 2 | 11
Haemorrhoids (Gastrointestinal disorders) | 7 | 6
Oral Candidiasis (Infections and infestations) | 2 | 11
Blood Alkaline Phosphatase Increased (Investigations) | 5 | 7
Amnesia (Nervous system disorders) | 4 | 7
Balance Disorder (Nervous system disorders) | 0 | 11
Glossodynia (Gastrointestinal disorders) | 4 | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 9
Paraesthesia (Nervous system disorders) | 2 | 9
Peripheral Motor Neuropathy (Nervous system disorders) | 3 | 8
Pyrexia (General disorders) | 3 | 7
Chills (General disorders) | 5 | 5
Hypoaesthesia (Nervous system disorders) | 3 | 6
Platelet Count Decreased (Investigations) | 6 | 4
Sinusitis (Infections and infestations) | 3 | 7
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 9
Blood Phosphorus Decreased (Investigations) | 4 | 5
Haemoglobin Decreased (Investigations) | 6 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Skin Discolouration (Skin and subcutaneous tissue disorders) | 7 | 2
White Blood Cell Count Decreased (Investigations) | 5 | 4
Disturbance in Attention (Nervous system disorders) | 4 | 4
Blood Calcium Decreased (Investigations) | 5 | 2
Neutrophil Count Decreased (Investigations) | 3 | 4
Non-Cardiac Chest Pain (General disorders) | 4 | 3
Dry Eye (Eye disorders) | 4 | 2
Proctalgia (Gastrointestinal disorders) | 3 | 3
Urinary Retention (Renal and urinary disorders) | 3 | 2
Blood Albumin Decreased (Investigations) | 3 | 1
Oedema (General disorders) | 3 | 0
Visual Field Defect (Nervous system disorders) | 3 | 12
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 3 | 7
Electrocardiogram T Wave Abnormal (Investigations) | 0 | 10
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes